CLINICAL TRIAL: NCT05693818
Title: A Multicenter, Single- Arm Study of Quantitative Assessment of Walking (Squawk) With the Canary canturioTM te (CTE) Tibial Extension
Brief Title: Quantitative Assessment of Walking (Squawk) With the Canary canturioTM te (CTE) Tibial Extension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Canary Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: POS-CTE-003
Record Dates: First submitted 2023-01-12; First posted 2023-01-23 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Arthritis Knee
Keywords: total knee arthroplasty; PersonaIQ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- PersonaIQ: Patients indicated for a PersonaIQ total knee arthroplasty
  Interventions: Other: Clinical Limping Evalution

INTERVENTIONS:
Other: Clinical Limping Evalution — Patients will be asked to perform a Clinical Limping Evaluation in the clinic during their post-operative follow-up visit. This will be performed in a controlled environment within the physician's clinic. Each patient will be asked to walk at their normal walking speed down a hallway for at least 7 consecutive steps and back toward the physician. Walking down the hallway and back is one walking trial. Each patient will be asked to perform 2 walking trials. The health care provider will assess the patient's limp using a 3-point Likert scale (0=No limp, 1=mild/moderate limp, 2=severe limp).
  If required, patients may use an assistive device and the type of device should be documented. If a patient requires assistance, only the minimum amount of assistance required for a patient to complete the task should be provided.
  Other Names: Limp Detection

SUMMARY:
The objective of this prospective study is to demonstrate accuracy of a limp detection model using a healthcare provider assessment as the non-reference standard.

DETAILED DESCRIPTION:
The primary endpoint of the study is limp severity at the 4-6 week office visit. At 4-6 weeks (+/- 3 days) post-surgery, the healthcare team will assess the patient's limp severity by visual observation on a 3-point Likert scale (0=No limp, 1=Mild/Moderate or 2=Severe).

ELIGIBILITY:
Inclusion Criteria:

* • Patient must be 18 years of age or older

  * Independent of study participation, patient is indicated for a commercially available PIQ TKA implant in accordance with product labeling
  * Patient must be willing and able to complete the protocol required follow-up
  * Patient has participated in the study-related informed consent process
  * Patient is willing and able to provide written Informed Consent by signing and dating the IRB approved informed consent

Exclusion Criteria:

* • Simultaneous bilateral TKA

  * Staged bilateral TKA less than 6 months from indexed procedure
  * Patient is a current alcohol or drug abuser
  * Patient is known to be pregnant, breastfeeding, or considered a member of a protected class (e.g., prisoner, mentally incompetent, etc.)
  * Patient has a psychiatric illness or cognitive deficit that will not allow proper informed consent and participation in follow-up program
  * Patient with mental or neurologic conditions who are unwilling or incapable of following postoperative care instructions
  * Patient with Neuropathic Arthropathy
  * Patient with any loss of musculature or neuromuscular disease that compromises the affected limb
  * Patients with known symptomatic foot, hip or spinal injuries and/or conditions that could affect gait

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients indicated for a commercially available PIQ TKA implant who meet the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Limp Severity | 4-6 wks+3 days weeks post TKA
  The primary endpoint of the study is limp severity at the 4-6 week office visit. At 4-6 weeks (+/- 3 days) post-surgery, the healthcare team will assess the patient's limp severity by visual observation on a 3-point Likert scale (0=No limp, 1=Mild/Moderate or 2=Severe).

SECONDARY OUTCOMES:
Test-retest reliability of the Canary Medical Limping Model (CMLM) score | 4-6 wks+3 days weeks post TKA
  Test-retest reliability of the CMLM score from day-to-day and week-to-week. (Specific days and weeks will be provided in the Statistical Analysis Plan.)
Positive Percent Agreement (PPA) of the CMLM with the healthcare team's assessment | 4-6 wks+3 days weeks post TKA
  Positive Percent Agreement (PPA)
Negative Percent Agreement (NPA) of the CMLM with the healthcare team's assessment | 4-6 wks+3 days weeks post TKA
  Negative Percent Agreement (NPA)
Knee Range of Motion | 4-6 wks+3 days weeks post TKA
  ROM will be measured by a goniometer
Numeric Pain Rating Scale | 4-6 wks+3 days weeks post TKA
  Subjective Pain Measurement
KOOS Jr | 4-6 wks+3 days weeks post TKA
  Patient Reported outcome
Limping Self Evaluation | 4-6 wks+3 days weeks post TKA
  Study participants will be asked the following question, "During the past week, have you been limping when walking, because of your knee?" The following answers will be allowed:
  * Rarely / never
  * Sometimes or just at first, after sitting for a long time
  * Often, not just at first
  * Most of the time
  * All of the time

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Orthopaedic & Neurosurgical Associates, Spartanburg, South Carolina, United States